CLINICAL TRIAL: NCT01213056
Title: Mindfulness-Based Cognitive Therapy for the Treatment of Chronic Headache Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09-0378
Record Dates: First submitted 2010-04-05; First posted 2010-10-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Headache; Pain
Keywords: Mindfulness Based Cognitive Therapy; Chronic Headache Pain; Randomized Controlled Trial.
MeSH Terms: conditions — Headache; Pain | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy * (MBCT) (Active Comparator): Mindfulness based cognitive therapy aimed to improve coping with, and managing chronic headache pain.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Delayed Treatment Control * (DT) (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Cognitive Behavioral (Active treatment condition)
  Arms: Mindfulness Based Cognitive Therapy * (MBCT)

SUMMARY:
The literature on the efficacy of Cognitive Behavioral Therapy (CBT) for the treatment of chronic pain is well established. Support for the efficacy of Mindfulness Based Stress Reduction (MBSR) and other mindfulness based treatments for chronic pain is building. Recently, research has demonstrated the efficacy of Mindfulness Based Cognitive Therapy (MBCT) in simultaneously addressing the outcome variables targeted by both CBT and mindfulness based treatment modalities. Although the efficacy of MBCT depression and for other populations has been investigated, there is no extant literature reporting on MBCT for chronic pain. The current application proposes to investigate the feasibility and efficacy of an MBCT protocoll adapted for chronic pain in a series of pilot groups with headache pain patients. We selected headache pain patients for this trial because headache pain is a common complaint in the general population, is the most frequently reported cause of pain in medical practice, and is one of the most disabling conditions for both genders combined. To examine the feasibility of the adapted protocol, the investigators will investigate a number of treatment related outcomes such as recruitment, completion, and drop out rates. Both primary and secondary outcome variables will be investigated to determine treatment efficacy.

This study will provide a research base examining the feasibility and efficacy of MBCT for pain. Results from this study will lay the foundation for future randomized controlled trials comparing MBCT to attention control, and future comparative effectiveness studies of MBCT and CBT.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy (CBT) is well established as an efficacious treatment for a wide variety of chronic pain conditions, including headache pain. A promising trend within the behavioral medicine field in recent years has been the integration of mindfulness into traditional treatment modalities and the development of innovative treatments based upon these principles. Mindfulness Based Stress Reduction (MBSR) maintains a patient-centered approach that focuses upon mindfulness meditation as the key mechanism to teach people how to cope with their pain, take better care of themselves, and to improve their overall quality of life. MBSR has successfully been utilized in a number of disorders including chronic pain 1,2,3 and in general medical populations 4 Mindfulness-Based Cognitive Therapy (MBCT),5 originally developed to target relapse prevention in major depression, is essentially a modification of MBSR to incorporate more traditional cognitive-behavioral interventions into the extant MBSR framework. Studies of MBCT support its efficacy in eliciting cognitive changes similar to those demonstrated in CBT, while still incorporating the more general salutary effects seen in MBSR,6,7,8,9,10While MBCT has been applied to other populations, there has been no published work to date adapting it to chronic pain patients. This is a surprising gap in the literature given the effectiveness of both CBT and mindfulness independently for chronic pain. Therefore, the present proposal seeks to begin to fill these gaps by testing the feasibility and efficacy of MBCT for chronic pain in a series of pilot groups.

Primary Specific Aims The proposed project is a feasibility study designed to test the MBCT protocol for chronic pain treatment and to provide pilot data to support subsequent research proposals to be submitted to the National Institutes of Health. In this initial trial the investigators will use patients with primary complaints of headache pain and treat them at a collaborating headache clinic. We selected this target population because headache pain is highly disabling and is the most common pain related complaint treated in medical practice. Furthermore, given the time frame of the study, it is more feasible to recruit patients where the PI has an established and ongoing collaborative relationship. The proposed project emphasizes the research area of health, medicine, and behavior.

Aim 1: To examine feasibility of the treatment, data will be collected regarding participant flow across each stage of the study design, including recruitment, participation, and drop-out rates, and percentage of sessions attended. Furthermore, pre-treatment expectations, post-treatment satisfaction, and global ratings of self-perceived improvement will be assessed.

Hypotheses: It is expected that the feasibility of MBCT, as measured by the above indicators, will be comparable to similar data for other psychosocial treatments for pain, such as CBT.

Aim 2: As an initial test of the efficacy of MBCT for chronic pain, the investigators will compare an immediate treatment condition to a delayed treatment (OT) control on pre- and post-intervention measures. Time constraints of the current project will necessitate follow-up assessment to be part of future proposals.

Hypotheses: Participants in the immediate treatment condition will obtain significantly greater pre-post treatment gains compared to OT on primary outcome measures of pain acceptance, pain catastrophizing, and pain interference; and secondary outcome measures of mindfulness, pain intensity, perceived disability, selfefficacy, quality of life, and depression.

Long-term objectives: Future projects will include a randomized controlled trial (RCT) comparing MBCT to an attention control condition (education support group), and eventually a comparative effectiveness stUdy of CBT vs. MBCT.

Innovative aspects of the proposed study: This is the first examination of MBCT for chronic pain, which incorporates specific components of mindfulness and cognitive behavioral therapy to form a comprehensive treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 pain days per month (for the past 3 months or more) due to migraine and/or tension-type headaches;
* Recent evaluation (within 6 months) of headaches by a physician, participants will also need to receive permission from their physician to take part in the study;
* Age of 19 years or older;
* Reading ability sufficient to comprehend self-monitoring forms;
* If currently using psychotropic or headache medications, use of these medications must have begun at least 4-weeks before treatment; and
* Agree to be videotaped during the group treatment sessions, although the video camera will be directed at the group leader, and not directed at the participant.

Exclusion Criteria:

* History of seizure or facial neuralgia, as these conditions might preclude the accurate diagnosis of headache;
* Significant cognitive impairment;
* History of schizophrenia, bipolar affective disorder or substance abuse as these conditions could result in a psychiatric emergency during treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Headache diary | 6 months
  Headache diary recordings of Headache Index, headache duration, headache frequency, and headache related disability.
  Pre-treatment, daily for two weeks prior to commencement of condition, daily during condition (i.e. both treatment and control condition participants complete the diary), post-treatment, 6-months follow-up.

SECONDARY OUTCOMES:
General Health Survey | 6 month follow-up
  General Health Survey Short-Form 36 (SF-36); The Migraine Disability Assessment (MIDAS); Beck Depression Inventory, Second Edition (BDI-II); Pain Catastrophizing Scale (PCS); Mindful Attention and Awareness Scale (MAAS); Chronic Pain Acceptance Questionnaire (CPAQ); Headache Management Self-Efficacy scale (HMSE); and Pain Appraisal Inventory (PAI).

CONTACTS AND LOCATIONS:
Overall Officials: Beverly E Thorn, Ph.D., Principal Investigator — University of Alabama, Tuscaloosa
Locations (1):
- UATuscaloosa, Tuscaloosa, Alabama, United States